CLINICAL TRIAL: NCT00330356
Title: Effects of Low Salt Diet Versus High Salt Diet on Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Wellcome Trust (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 074825/Z/04/Z
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Last update posted 2006-05-26 (Estimated); Status verified 2006-04

CONDITIONS: Hypertension
Keywords: Dietary Salt; Blood Pressure; Normotensives
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Behavioral: Low Salt Diet versus High salt diet

SUMMARY:
High blood pressure is a global public health problem in developed and developing countries including Pakistan. Various studies conducted around the world have linked salt intake to variation in the blood pressure.However, definite conclusions are lacking and the exact role of dietary salt in salt-blood pressure relationship remains controversial.

While clinical practice guidelines recommend dietary salt restriction for lowering blood pressure, the relationship of salt with blood pressure has not been tested in the Pakistani population. Therefore, the efficacy of dietary salt restriction on blood pressure of this population remains to be determined. The study aims to determine the relationship between dietary salt intake and blood pressure in Pakistani population. It is hypothesized that alteration in the dietary salt intake demonstrates significant changes in the Systolic BP.

DETAILED DESCRIPTION:
High blood pressure is a global public health problem in developed and developing countries including Pakistan. Various studies conducted around the world have linked salt intake to variation in the blood pressure.However, definite conclusions are lacking and the exact role of dietary salt in salt-blood pressure relationship remains controversial.

While clinical practice guidelines recommend dietary salt restriction for lowering blood pressure, the relationship of salt with blood pressure has not been tested in the Pakistani population. Therefore, the efficacy of dietary salt restriction on blood pressure of this population remains to be determined.

Objectives:

* To assess the effects of low salt diet versus high salt diet on blood pressure in normotensive adults aged 40 years or above in Karachi, Pakistan
* To estimate the prevalence of salt sensitivity and salt resistance in normotensive adults aged 40 years or above in Karachi, Pakistan

Study Design:

The proposed study is a prospective, randomized, crossover, open label evaluation trial.

Study Population & setting:

For the proposed study, subjects age 40 or over without hypertension and fulfilling the eligibility criteria will be randomly selected.Informed consent will be obtained.

Each participant would then be randomized to either low salt (sodium 20mmol/day) or high salt diet (sodium 220mmol/day) for one week, with a washout period of regular diet for one week, and the reverse of initial randomization for another week.

Blood pressure at baseline and at the end of each intervention week would be measured using a calibrated automated device in the sitting position from the right arm after 5 minutes of rest using an appropriate sized cuff. Three consecutive readings with an interval of 05 minutes will be taken and the mean of the final two blood pressure readings will be used in the analysis. Compliance to the diet will be confirmed by measuring 24-hour urinary sodium and urinary creatinine throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 40 years and above

  * With systolic BP <140 and diastolic < 90 mmHg
  * Not receiving pharmacological antihypertensive medications

Exclusion Criteria:

* Subjects with following conditions would be excluded:

  * Diabetes mellitus (positive history of diabetes or fasting blood sugar ≥ 126 mg/dl)
  * Renal insufficiency (serum creatinine of 1.4 mg/dl or above)
  * Pregnant or lactating women

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-09; Study Completion 2006-04

PRIMARY OUTCOMES:
Difference in mean systolic blood pressure (SBP) between completion of the high salt phase compared with the low salt phase.

SECONDARY OUTCOMES:
Salt Sensitivity defined as an increase in SBP of at least 8 mmHg at the end of high salt phase compared with the end of low salt phase.
Salt Resistance would be defined as those with rise of < 4 mm Hg of SBP at the end of high salt phase compared with the end of low salt phase.

CONTACTS AND LOCATIONS:
Overall Officials: Tazeen H Jafar, MD, MPH, Study Director — Aga Khan University; Saleem Jessani, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Jessani S, Hatcher J, Chaturvedi N, Jafar TH. Effect of low vs. high dietary sodium on blood pressure levels in a normotensive Indo-Asian population. Am J Hypertens. 2008 Nov;21(11):1238-44. doi: 10.1038/ajh.2008.256. Epub 2008 Sep 4. PMID 18772855